CLINICAL TRIAL: NCT02161146
Title: AGN-229666 Ophthalmic Solution in Japanese Patients With Allergic Conjunctivitis
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Allergan (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: 229666-006
Record Dates: First submitted 2014-06-09; First posted 2014-06-11 (Estimated); Results first posted 2016-03-07 (Estimated); Last update posted 2019-04-17 (Actual); Status verified 2019-04

CONDITIONS: Conjunctivitis, Allergic
MeSH Terms: conditions — Conjunctivitis, Allergic | interventions — Olopatadine Hydrochloride

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (5):
- AGN-229666 (Experimental): One drop of AGN-229666 in each eye on Days 1 and 15.
  Interventions: Drug: AGN-229666
- Vehicle (Placebo Comparator): One drop of Vehicle to AGN-229666 in each eye on Days 1 and 15.
  Interventions: Drug: Vehicle to AGN-229666
- Olopatadine (Active Comparator): One drop of olopatadine in each eye on Days 1 and 15.
  Interventions: Drug: Olopatadine
- AGN-229666/Olopatadine (Other): One drop of AGN-229666 in one eye and one drop of olopatadine in the other eye on Days 1 and 15.
  Interventions: Drug: AGN-229666; Drug: Olopatadine
- AGN-229666/Vehicle (Other): One drop of AGN-229666 in one eye and one drop of Vehicle to AGN-229666 in the other eye on Days 1 and 15.
  Interventions: Drug: AGN-229666; Drug: Vehicle to AGN-229666

INTERVENTIONS:
Drug: AGN-229666 — One drop of AGN-229666 in the eye on Days 1 and 15.
  Arms: AGN-229666; AGN-229666/Olopatadine; AGN-229666/Vehicle
Drug: Vehicle to AGN-229666 — One drop of Vehicle to AGN-229666 in the eye on Days 1 and 15.
  Arms: AGN-229666/Vehicle; Vehicle
Drug: Olopatadine — One drop of olopatadine in the eye on Days 1 and 15.
  Other Names: Patanol®
  Arms: AGN-229666/Olopatadine; Olopatadine

SUMMARY:
This study will evaluate the safety and efficacy of AGN-229666 for the prevention of allergen-mediated conjunctivitis.

ELIGIBILITY:
Inclusion Criteria:

-Japanese patients living in Japan with a history of allergic conjunctivitis.

Exclusion Criteria:

* Presence of active eye infection (bacterial, viral, or fungal)
* History of an eye herpetic infection.

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 240 (Actual)
Dates: Start 2014-06-04 (Actual); Primary Completion 2014-12-20 (Actual); Study Completion 2014-12-20 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Allergan
Locations (1):
- Tokyo, Japan

REFERENCES:
- [Background] Nakatani H, Gomes P, Bradford R, Guo Q, Safyan E, Hollander DA. Alcaftadine 0.25% versus Olopatadine 0.1% in Preventing Cedar Pollen Allergic Conjunctivitis in Japan: A Randomized Study. Ocul Immunol Inflamm. 2019;27(4):622-631. doi: 10.1080/09273948.2018.1432764. Epub 2018 Mar 15. PMID 29543548

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | AGN-229666 | Vehicle | Olopatadine | AGN-229666/Olopatadine | AGN-229666/Vehicle
Started | 47 | 47 | 49 | 48 | 49
Completed | 46 | 43 | 49 | 45 | 48
Not Completed | 1 | 4 | 0 | 3 | 1
Not completed — Adverse Event | 1 | 1 | 0 | 1 | 0
Not completed — Lost to Follow-up | 0 | 1 | 0 | 0 | 0
Not completed — Personal Reasons | 0 | 1 | 0 | 2 | 1
Not completed — Other Miscellaneous Reasons | 0 | 1 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | AGN-229666 | Vehicle | Olopatadine | AGN-229666/Olopatadine | AGN-229666/Vehicle | Total
Number analyzed (Participants) | 47 | 47 | 49 | 48 | 49 | 240
Age, Customized [Number; unit: participants]
  20 to 30 years | 22 | 15 | 16 | 21 | 20 | 94
  >30 to 40 years | 9 | 12 | 7 | 7 | 7 | 42
  >40 years | 16 | 20 | 26 | 20 | 22 | 104
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 17 | 22 | 24 | 19 | 26 | 108
  Male | 30 | 25 | 25 | 29 | 23 | 132

OUTCOME MEASURES:

1. Primary Outcome: Ocular Itching Score
Description: Ocular itching was assessed by the participant 8 hours after AGN-229666 and vehicle administration and 4 hours after olopatadine administration, 5 minutes post allergen challenge using a 0 to 4 scale with 0.5 grade increments where: 0=none (no itching) to 4.0=incapacitating itch with an irresistible urge to rub (worst). Data from Days 1 and 15 were pooled together and averaged.
Time Frame: Days 1 and 15
Population: Participants from the Intent-to-Treat Population, all randomized participants, with data of treated eyes available for analysis.
Measure: Mean (Standard Deviation); unit: score on a scale
Units Other Than Participants: Eyes
Groups:
- Vehicle: One drop of Vehicle to AGN-229666 in the eye on Days 1 and 15.
Arm/Group | AGN-229666 | Vehicle | Olopatadine
Number analyzed (Participants) | 144 | 96 | 97
Number analyzed (Eyes) | 186 | 136 | 145
score on a scale | 0.33 (0.523) | 1.48 (0.904) | 0.29 (0.411)

2. Secondary Outcome: Conjunctival Hyperemia Score
Description: Hyperemia is the engorgement of the blood vessels (redness) of the eye. Ocular hyperemia was evaluated by the investigator 8 hours after AGN-229666 and vehicle administration and 4 hours after olopatadine administration, 15 minutes post allergen challenge using a 0 to 4 scale with 0.5 grade increments where: 0=none (no hyperemia) to 4.0=extremely severe (large, numerous dilated blood vessels characterized by severe deep red color). Data from Days 1 and 15 were pooled together and averaged.
Time Frame: Days 1 and 15
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: score on a scale
Units Other Than Participants: Eyes
Arm/Group | AGN-229666 | Vehicle | Olopatadine
Number analyzed (Participants) | 144 | 96 | 97
Number analyzed (Eyes) | 186 | 136 | 145
score on a scale | 1.15 (0.771) | 1.61 (0.820) | 1.34 (0.849)

ADVERSE EVENTS:
Arm/Group | AGN-229666 | Vehicle | Olopatadine | AGN-229666/Olopatadine | AGN-229666/Vehicle
Serious Adverse Events (participants affected / at risk) | 0/47 | 0/47 | 0/49 | 0/48 | 0/49
Other Adverse Events (participants affected / at risk) | 4/47 | 10/47 | 6/49 | 3/48 | 5/49
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | AGN-229666 (N=47) | Vehicle (N=47) | Olopatadine (N=49) | AGN-229666/Olopatadine (N=48) | AGN-229666/Vehicle (N=49)
Nasopharyngitis (Infections and infestations) | 3 | 1 | 1 | 0 | 2
Oropharyngeal discomfort (Respiratory, thoracic and mediastinal disorders) | 1 | 6 | 3 | 2 | 1
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 1 | 3 | 2 | 1 | 2
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 1 | 3 | 2 | 0 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
A disclosure restriction on the PI is that the sponsor can review results communications prior to public release and can embargo communications regarding trial results for a period that is less than or equal to 90 days from the time submitted to the sponsor for review. The sponsor cannot require changes to the communication and cannot extend the embargo.